CLINICAL TRIAL: NCT06296836
Title: Effect of Continuing Versus Holding Metformin During Hospitalizations to Internal Medicine on Glucose Control, Acidosis, Abdominal Symptoms, Length of Stay, and Mortality.
Brief Title: Effect of Continuing Versus Holding Metformin During Hospitalizations.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-001
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, prospective trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin continuation (Active Comparator): Continuation of home metformin regimen during hospitalization to an internal medicine service
  Interventions: Drug: Metformin
- Metformin discontinuation (No Intervention): Holding home metformin regimen during hospitalization to an internal medicine service

INTERVENTIONS:
Drug: Metformin — Continuation of home metformin
  Other Names: Glucophage
  Arms: Metformin continuation

SUMMARY:
A randomized study of continuing versus holding metformin during hospitalizations to internal medicine services to determine the effects on glucose control, acidosis, abdominal symptoms, length of stay, and mortality.

DETAILED DESCRIPTION:
The purpose of this study is to determine what the effects of the routine practice of holding metformin in hospitalized patients with type 2 diabetes are on outcomes.

The objectives of this study are to determine how holding versus continuing metformin during hospitalization to an internal medicine service affects the incidences of lactic acidosis, mean anion gap, mean glucose levels, low and very high blood sugars, GI effects after discharge, lack of continuation of metformin upon discharge, mean glucose levels, lengths of stay, and 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Admitted to an internal medicine service.
* On Metformin prior to admission.

Exclusion Criteria:

* Inability to take oral medications
* eGFR < 30 ml/min/1.73 m2
* Dialysis
* Current Acidosis (pH < 7.35) including diabetic ketoacidosis
* Child-Turcotte-Pugh class C hepatic cirrhosis
* Acute Decompensated Heart Failure
* Cognitively impaired and/or unable to consent
* Lack of or unwillingness to share contact information
* Pregnant women

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean glucose levels | During hospitalization
  Average of daily glucose levels during hospitalization

SECONDARY OUTCOMES:
Incidence of hyperglycemia greater than 300 mg/dl. | During hospitalization
  Glucose > 300
Incidence of hypoglycemia (Glu = 54 - 70). | During hospitalization
  Glu = 54 - 70
Incidence of moderate hypoglycemia (Glu < 54) | During hospitalization
  Glu < 54
Incidence of severe hypoglycemia (Glu < 54 with symptoms) | During hospitalization
  Glu < 54 with symptoms
Mean lactic acid levels. | During hospitalization
  Mean lactic acid levels
Incidence of lactic acid levels greater than 2.0. | During hospitalization
  Lactic acid > 2.0
Mean anion gap. | During hospitalization
  Mean anion gap, a calculated value
Incidence of anion gap > 11 | During hospitalization
  Anion Gap > 11
Incidence of elevated lactic acid level or anion gap. | During hospitalization
  Lactic acid > 2.0 or Anion Gap > 11
Incidence of inadvertently not continuing metformin on discharge | At discharge
  Transitions of care
GI adverse effects | Within 3 days of discharge
  GI side effects after discharge
Mortality | 30 +/- 3 days after discharge
  Mortality as determined via chart search and follow up phone call

OTHER OUTCOMES:
Mean glucose levels while receiving metformin in the continuation arm and while not receiving metformin in the discontinuation arm | During hospitalization
  Mean daily glucose levels will only be included for the days in which the subjects received or did not receive metformin as per their assigned arm.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No